CLINICAL TRIAL: NCT02473692
Title: Examining Feasibility and Effectiveness of an Internet-based Intervention for Facilitating Migraine Medication Adherence and Optimizing Medication Use
Brief Title: Facilitating Migraine Medication Adherence and Optimizing Medication Use
Status: Withdrawn | Type: Observational
Why Stopped: Delays in start date led to termination of the study prior to recruitment of participants.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MK-0974
Record Dates: First submitted 2015-05-29; First posted 2015-06-16 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-08

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online MigraineTreatment Optimization: After providing informed consent, participants will complete a series of questionnaires related to their headaches and medication beliefs. After completion, they will have full access to an informational website including access to text-based supplemental materials pertaining to headache and headache treatment, and a series of videos designed specifically for this trial. Participants will be asked to watch seven videos of approximately four-minute length each and to complete a post-assessment question following the completion of each of the first 6 videos. The total time required to complete all study activities will be approximately one hour.
  Interventions: Other: Online Migraine Treatment Optimization

INTERVENTIONS:
Other: Online Migraine Treatment Optimization — The educational videos entail a young woman (i.e., an actress) describing her experiences in managing her headaches. The informational content of the videos is organized into 7 content areas that present a wealth of information in an entertaining way:
  1. Introduction to the series
  2. Getting to know migraine
  3. Making the most of your medical care
  4. Partnering with your doctor
  5. Best use of migraine medication
  6. Keeping tabs on your migraine
  7. Take home message (summary)

SUMMARY:
The present research will pilot-test a new state-of-the-art Internet-based intervention targeting adherence facilitation and optimization of medication use, and will be evaluated to assess its utility in facilitating adherence and optimization of medication use for acute migraine pharmacotherapy. This is not an interventional study and will instead be an observational assessment of the feasibility of an online program (a proof-of-concept study). The two principal objectives of this study include: (a) examination of the feasibility and user usage patterns of an Internet-based intervention designed to potentially enhance adherence to medication use recommendations, and (b) determination of the efficacy of the Internet-based intervention in potentially increasing knowledge of abortive medication-use guidelines and in improving adherence to those guidelines. To meet the objectives of this study, a website has been specifically developed including a series of supplemental text-based headache materials and a series of videos based social learning theory and modeling principles (as opposed to the stereotypical 'talking-heads' mode of information delivery).

DETAILED DESCRIPTION:
Objective 1. To examine the feasibility and user usage patterns/demand of an online intervention designed to enhance adherence and optimize abortive medication-use for migraineurs.

Goal 1: To evaluate the practical utility of an Internet-based user environment to host an intervention designed to increase knowledge of and facilitate adherence and optimize abortive medication use.

Hypothesis 1A: That an Internet-based user environment can be appropriately suited to deliver an adherence intervention that, in turn, could be made widely accessible and readily employed.

Hypothesis 1B: That a high proportion of patients referred to the adherence facilitation Web site will actually visit and make use of the adherence intervention Web site.

Hypothesis 1C: That once the Web-based intervention is initiated, a low attrition rate will be observed and the majority of patients will complete the intervention.

Objective 2. To examine the efficacy of an online adherence facilitation and medication optimization intervention in increasing knowledge of optimal abortive medication-use.

Goal 2: To conduct a pilot trial examining the efficacy of an adherence and medication optimization intervention for improving knowledge and medication-use behavior in a wide range of migraine sufferers.

Hypothesis 2A: That patients who complete the Web-based intervention will demonstrate improved knowledge of optimal abortive medication strategies at post-treatment and this knowledge will be maintained at follow-up.

Hypothesis 2B: That patients who complete the Web-based intervention will report improved abortive medication use strategies at post-treatment and this behavior change will be maintained at follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Adults >= 18 year-old
2. Any self-reported headache disorder, from any etiology ( > 5 attacks, lifetime)
3. Self-reported use of any headache abortive treatment:

   * Over the counter (e.g., Ibuprofen, naproxen sodium, Excedrin, etc.)
   * Prescription (Triptans, CGRP antagonist, Ibuprofen, etc.)

Exclusion Criteria

1. Inability to read and write English (the questionnaires are exclusively in English)
2. Inability to accurately complete questionnaire or provide informed consent: (e.g., Florid psychosis, Current intoxication)
3. No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll N = 300 participants. The proposed study is primarily powered to estimate the rate at which headache patients will likely seek out the Web site within a desired precision range (i.e., Hypothesis 1A). This sample size will allow the characterization of the various event rates within a precise range. For example, this sample size would allow a precision of +/- 5% around most event rates (i.e., use rates, attrition rates, etc.). Finally, even with a large attrition rate (i.e., 50%) the proposed sample size will allow the detection of even small changes (e.g., d = 0.20) in the adherence measures (assuming adequate reliability, and a modest correlation between measurement occasions).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by the practical utility of an Internet-based user environment to host an intervention designed to increase knowledge of and facilitate adherence to abortive medication use guidelines. | Post-intervention, at the end of the 1 week study period
  Feasibility will be demonstrated based on the number of participants who complete the online videos.

SECONDARY OUTCOMES:
Attrition assessed by the rate of attrition from the study, determined based upon the number of enrolled participants who do not complete the online video portion. | Post-intervention, at the end of the 1 week study period
  Attrition assessed by the rate of attrition from the study, determined based upon the number of enrolled participants who do not complete the online video portion.

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Penzien, PhD, Principal Investigator — WakeForest School of Medicine